CLINICAL TRIAL: NCT01097278
Title: Phase IIB Randomized Controlled Biomarker Modulation Study of Vitamin D in Premenopausal Women at High Risk for Breast Cancer
Brief Title: S0812 High Dose Cholecalciferol in Premenopausal Women at High-Risk for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S0812; S0812 (Other: SWOG); U10CA037429 (NIH); NCI-2011-02032 (Other: NCI)
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: brca1 Mutation Carrier; brca2 Mutation Carrier; Breast Cancer
Keywords: breast cancer; ductal breast carcinoma in situ; lobular breast carcinoma in situ; BRCA1 mutation carrier; BRCA2 mutation carrier
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Randomized Phase 2 study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Participants receive oral cholecalciferol once weekly and oral vitamin D once daily. Treatment repeats for 12 months in the absence of evidence of cancer or unacceptable toxicity.
  Interventions: Dietary Supplement: cholecalciferol
- Arm II (Active Comparator): Participants receive oral placebo once weekly and oral vitamin D once daily. Treatment repeats for 12 months in the absence of evidence of cancer or unacceptable toxicity.
  Interventions: Dietary Supplement: cholecalciferol; Other: placebo

INTERVENTIONS:
Dietary Supplement: cholecalciferol — Given orally
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Cholecalciferol may prevent breast cancer in premenopausal women.

PURPOSE: This randomized phase II trial is studying how well cholecalciferol works in preventing breast cancer in premenopausal women.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess whether mammographic density is reduced in premenopausal women at high risk of breast cancer taking high-dose vitamin D3 (oral cholecalciferol 20,000 IU weekly) vs placebo for 1 year.
* To assess whether proliferation as measured by Ki-67 staining of breast epithelial cells is reduced in women receiving these treatments.
* To explore the difference in the expression of other biomarkers (including cleaved caspase-3 [apoptosis marker], ER, vitamin D receptor [VDR], and 1α-hydroxylase) in breast tissue obtained from these women.
* To assess whether parathyroid hormone, IGF-1, IGFBP-3, 25(OH)D, and 1,25(OH)D serum levels are altered in these women at baseline and at 6 and 12 months.
* To explore whether a change in mammographic density correlates with polymorphisms in the VDR gene.
* To assess other sources of vitamin D (sunlight exposure, diet) in these women using a validated questionnaire administered at baseline and at 12 and 24 months.
* To collect and bank serum, plasma, and breast tissue from these women before and after a 1-year intervention with vitamin D for future biomarker analysis.
* To assess the toxicity of high-dose cholecalciferol compared to placebo in this setting.

OUTLINE: This is a multicenter study. Participants are stratified according to baseline serum 25(OH)D level (< 20 ng/mL vs 20-32 ng/mL or < 50 nmol/L vs 50-80 nmol/L), baseline mammographic density (11-50% vs > 50%), and designated biopsy site (yes vs no). Participants are randomized to 1 of 2 treatment arms.

* Arm I: Participants receive oral cholecalciferol once weekly and oral vitamin D once daily. Treatment repeats for 12 months in the absence of evidence of cancer or unacceptable toxicity.
* Arm II: Participants receive oral placebo once weekly and oral vitamin D once daily. Treatment repeats for 12 months in the absence of evidence of cancer or unacceptable toxicity.

Blood samples are collected at baseline and periodically thereafter for biomarkers and 25(OH)D level. Participants undergo a mammogram at baseline and at 12 months. Participants may also undergo random core-needle breast biopsy at baseline and at 12 months.

Participants complete a questionnaire at baseline and at 12 and 24 months.

After completion of study therapy, participants are followed up at 1 and 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At an elevated risk of breast cancer by at least one of the following criteria:

  * Diagnosis of ADH, ALH, lobular carcinoma in situ (LCIS) or resected ductal carcinoma in situ (DCIS) or small invasive breast cancers (pTmi or pT1a N0) if no pior RT, tamoxifen, or systemic breast cancer treatment within 28 days prior to registration OR diagnosis of resected Stage I (T1b-c N0-N1mi) through Stage II breast cancer for which the participant has been disease-free for at least 5 years and has completed all adjuvant treatment OR
  * A known* deleterious mutation in BRCA1, BRCA2, PTEN, or TP53 NOTE: *The participant must be a documented carrier to meet this criterion. If there is a known mutation in a hereditary breast cancer susceptibility gene in a participant's family member, the participant herself must have undergone genetic testing as per NCCN clinical guidelines to be eligible per this criterion.
  * Modified Gail Model/CARE model** risk at 5 years ≥ 1.67% or lifetime risk ≥ 20% by Claus, BRCAPro, Tyrer-Cuzick or IBIS models OR
  * Mammographic density ≥ 50% (heterogenously dense) NOTE: **Risk models are to be used only if there is no known previous diagnosis of resected DCIS or LCIS and there is no known deleterious mutation in BRCA1, BRCA2, PTEN, or TP53.
* At least one breast available for imaging and biopsy (a previously irradiated breast [i.e., for resected DCIS] is not evaluable for breast imaging or biopsy)
* Baseline mammogram (performed within 10 days after starting their last menstrual period on a digital mammography machine) that shows either normal or benign findings

  * Baseline mammographic density > 10% based upon the classification system (2 = 11-50%, "scattered fibroglandular densities"; 3 = 51-75%, "heterogeneously dense"; 4 = >75, "extremely dense". Women with a baseline mammographic density of ≤ 10% (1 = ≤ 10% breasts are almost entirely fat)will not be eligible.

PATIENT CHARACTERISTICS:

* Premenopausal, defined as ≥ 1 of the following criteria:

  * Less than 6 months since the last menstrual period, no prior bilateral oophorectomy, and no use of hormone-replacement therapy
  * Has undergone a prior hysterectomy but no prior bilateral oophorectomy AND follicle-stimulating hormone values measured within the past 28 days are consistent with the normal values for the premenopausal state
* Zubrod performance status 0-1
* Serum creatinine ≤ upper limit of normal (ULN)
* Serum calcium or corrected calcium ≤ ULN
* Spot urine calcium:creatinine ratio < 0.37 mg/dL
* INR ≤ 1.5 times ULN+
* PT and PTT ≤ ULN*
* Baseline serum 25(OH)D level ≤ 32 ng/mL (or 80 nmol/L)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other prior malignancy except for the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Adequately treated stage I or II (including resected Stage I, T1b-c N0-N1mi through Stage II breast cancer) from which the participant is currently in complete remission
  * Any other cancer (including contralateral breast) for which the participant has been disease-free for ≥ 5 years
* No history of kidney stones
* No medical conditions requiring calcium or vitamin D supplementation (i.e., osteoporosis)
* No known hypersensitivity to vitamin D
* No known allergy to soy NOTE: +For patients undergoing breast biopsy.

PRIOR CONCURRENT THERAPY:

* Prior breast reduction surgery allowed

  * No bilateral breast implants
* More than 1 month since prior surgery or radiotherapy to the breast for resected DCIS
* At least 28 days since prior tamoxifen
* Prior anticoagulant therapy allowed provided it is discontinued ≥ 7 days before breast biopsy
* No concurrent calcium or additional vitamin D supplements

  * Concurrent multivitamins allowed provided that the dose of vitamin D in the multivitamin does not exceed 400 IU daily
* No concurrent participation in any other clinical trial for the treatment or prevention of cancer unless the participant is no longer receiving the intervention and is in the follow-up phase only (participants must not join such a trial while participating in this study)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 208 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in mammographic density at 12 months compared to baseline | 12 months

SECONDARY OUTCOMES:
Ki-67 as assessed in tissue obtained in breast biopsies at baseline and at 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Katherine D. Crew, MD, MS, Principal Investigator — Columbia University
Locations (360):
- United States (360):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Providence Hospital, Mobile, Alabama
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Highlands Oncology Group-Rogers, Rogers, Arkansas
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Huntington Memorial Hospital, Pasadena, California
  - East Bay Medical Oncology Hematology Medical Associates Inc-Pleasant Hill, Pleasant Hill, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Breastlink Medical Group Inc, Santa Ana, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Greenwich Hospital, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Florida Hospital Orlando, Orlando, Florida
  - Martin Medical Center, Stuart, Florida
  - Robert and Carol Weissman Cancer Center at Martin Health, Stuart, Florida
  - Martin Hospital South, Stuart, Florida
  - Dekalb Medical Center, Decatur, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Oncare Hawaii Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg Cottage Plaza Office, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Mid-Illinois Hematology Oncology Associates Limited, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Cancer Care Partners LLC, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baptist Health Corbin, Corbin, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Hematology/Oncology Clinic LLP, Baton Rouge, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Steward Saint Elizabeth's Medical Center, Brighton, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Botsford General Hospital, Farmington, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mid-Michigan Medical Center - Midland, Midland, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center-Carrie J Babb Cancer Center, Bolivar, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Winthrop University Hospital, Mineola, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Hematology Oncology Associates of Central New York-Rome, Rome, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Hematology Oncology Associates of Central New York-Onondaga Hill, Syracuse, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Park Ridge Hospital Breast Health Center, Hendersonville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Novant Health Cancer Specialists-Matthews, Matthews, North Carolina
  - Lake Norman Hematology Oncology Specialists-Mooresville, Mooresville, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Trinity Cancer Care Center, Minot, North Dakota
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Western Oncology Research Consortium, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Carolina Blood and Cancer Care Associates PA, Rock Hill, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Texas Tech University Health Science Center-Amarillo, Amarillo, Texas
  - Baylor University Medical Center, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - The Methodist Hospital System, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - EvergreenHealth Medical Center, Kirkland, Washington
  - Virginia Mason CCOP, Seattle, Washington
  - Pacific Medical Center-First Hill, Seattle, Washington
  - Rockwood Clinic, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Princeton Community Hospital, Princeton, West Virginia
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming